CLINICAL TRIAL: NCT00750646
Title: The Relationship Between Glaucoma Medication Self-Efficacy, Outcome Expectations, Eye Drop Tech., Adherence and IOP.
Brief Title: Observational Study of How Patients Take Eye Drops
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Robin, Alan L., M.D. (Individual)
Collaborators: Alcon Research (Industry)
Responsible Party: Alan L. Robin, Glaucoma Specialists
Other Study IDs: SI-08-54
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Last update posted 2008-09-10 (Estimated); Status verified 2008-09

CONDITIONS: Glaucoma
Keywords: compliance; eye drop administration; MEMS; adherence
MeSH Terms: conditions — Glaucoma; Patient Compliance | interventions — Micro-Electrical-Mechanical Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- A: Subject's adherence to prescribed therapy will be monitored with an electronic compliance device.
  Interventions: Device: MEMS cap

INTERVENTIONS:
Device: MEMS cap — The Medication Event Monitoring System will be used to assess the level of subject adherence to recommended topical eye drop therapy.
  Other Names: MEMS

SUMMARY:
This study is interested in monitoring how patients take eye drops, both through video-recordings and adherence monitoring, as well as their perceptions about their eye medications; including the dosing schedules, instillation techniques and effect on their disease.

ELIGIBILITY:
Inclusion Criteria:

* >18 year old
* currently taking 1 or more hypotensive topical eye drops takes drops in the right eye for more than 6 months expect to continue drop use for the next 3 months
* subjects instill their own eye drops
* subject is able to take HVF tests
* subject will expect to complete the 3 months enrollment period

Exclusion Criteria:

* unable/unwilling to instill own medications
* eye drops are discontinued
* unable to take HVF test
* unable to complete follow-up
* investigators discontinue subject for safety reasons
* not using drops in left eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be enrolled for a single site, private practice.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-03 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Medication adherence measured by MEMS caps | 3 months
Eye drop technique measured by video evaluation | 1 time observation

SECONDARY OUTCOMES:
Medication adherence measured by self-report | 3 months
Severity of VF damage | 1 test date
Intraocular pressure readings | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Stone, OD, Principal Investigator — Glaucoma Experts; Alan L Robin, MD, Principal Investigator — Glaucoma Specialists; Colleen K Protzko, Study Director — Glaucoma Specialists
Locations (1):
- Glaucoma Specialists, Baltimore, Maryland, United States